CLINICAL TRIAL: NCT00857519
Title: Intra-arterial (Ophthalmic Artery) Chemotherapy for Retinoblastoma
Brief Title: A Study of the Effectiveness of a Local Injection of Chemotherapy for Retinoblastoma
Acronym: IAC-RB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Carol L Shields, Carol L. Shields, MD Co-Director, Ocular Onology Service, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-885
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Retinoblastoma
Keywords: retinoblastoma; Intraarterial; Chemotherapy; Melphalan; Carboplatin
MeSH Terms: conditions — Retinoblastoma | interventions — Melphalan; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy (Experimental): Chemotherapy using Melphalan, Carboplatin.
  Interventions: Drug: Melphalan, Carboplatin

INTERVENTIONS:
Drug: Melphalan, Carboplatin — Intra-arterial chemotherapy.
  Other Names: ALKERAN,PARAPLATIN

SUMMARY:
Over the past 15 years, intravenous chemotherapy has become the most popular conservative (eye-saving) method for retinoblastoma treatment because it is often effective and usually safe. In recent years, there has been much interest in providing highly focused (focal) chemotherapy to a diseased organ including the liver, brain, and eye. With focused chemotherapy, the chemotherapy drugs are injected directly into the ophthalmic artery (the artery that supplies blood to the eye). A benefit of focal chemotherapy delivery is that it decreases the chance of toxicity to other organs such as bone marrow suppression (causing low blood counts) and the development of other cancers in the future.

DETAILED DESCRIPTION:
The management of retinoblastoma includes systemic chemotherapy (carboplatin, etoposide, and vincristine), thermotherapy, cryotherapy (freezing treatment), laser photocoagulation, plaque radiotherapy, external beam radiotherapy, and enucleation. The treatment is tailored to each individual case. Over the past 15 years, intravenous chemotherapy has risen as the most popular conservative (eye-saving) method for retinoblastoma management because it is effective and safe. In recent years, there has been keen interest in providing chemotherapy more focally to a diseased organ including the liver, brain, and eye. The benefit of focal chemotherapy delivery is to avoid toxicity to other organs and this toxicity includes the risk of future cancers.

ELIGIBILITY:
Inclusion Criteria:

* Advanced retinoblastoma in one or both eyes
* Recurrent retinoblastoma after failure of previous treatment
* No age limit (usually kids presenting with retinoblastoma present in the 1st two decades of life)
* Judged by principal investigator to be medically and physically able to undergo the procedure

Exclusion Criteria:

* Recurrent retinoblastoma which is treatable with other conservative measures
* Invasive retinoblastoma (retinoblastoma that has grown locally outside of the eye, for example, into the bone around the eye)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Tumor control | after 5 cycles of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Shields, MD, Principal Investigator — Oncology Service, Wills Eye Institute
Locations (1):
- Oncology Service, Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuncer S, Balci O, Tanyildiz B, Kebudi R, Shields CL. Intravitreal Lower-Dose (20 microg) Melphalan for Persistent or Recurrent Retinoblastoma Vitreous Seeds. Ophthalmic Surg Lasers Imaging Retina. 2015 Oct;46(9):942-8. doi: 10.3928/23258160-20151008-07. PMID 26469234
- [Background] Shields CL, Manjandavida FP, Arepalli S, Kaliki S, Lally SE, Shields JA. Intravitreal melphalan for persistent or recurrent retinoblastoma vitreous seeds: preliminary results. JAMA Ophthalmol. 2014 Mar;132(3):319-25. doi: 10.1001/jamaophthalmol.2013.7666. PMID 24407202